CLINICAL TRIAL: NCT01849562
Title: A Phase 2a Trial to Evaluate the Safety, Tolerability, and Efficacy of 12 Weeks of Sovaprevir, ACH-0143102 and Ribavirin in Treatment-Naive Subjects With Chronic Hepatitis C Genotype-1 Viral Infection
Brief Title: Safety, Tolerability, and Efficacy of 12-weeks of Sovaprevir, ACH-3102, and Ribavirin in Treatment-naive GT-1 HCV Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH102-007
Record Dates: First submitted 2013-04-18; First posted 2013-05-08 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic Hepatitis C; Genotype 1; Hepatitis C; Liver Diseases; Hepatitis; Ribavirin; Antiviral Agents; Anti-infective Agents; Protease Inhibitors; NS5a Inhibitors; Viral
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Liver Diseases; Hepatitis | interventions — odalasvir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sovaprevir 200 milligrams (mg), ACH-3102 150/50 mg, RBV 1000-1200 mg (Active Comparator): Sovaprevir 200 mg once daily (qd) + ACH-3102 150 mg loading dose on Day 1, followed by 50 mg qd + RBV weight-based 1000-1200 mg qd for 12 weeks.
  Interventions: Drug: Sovaprevir; Drug: ACH-3102; Drug: Ribavirin
- Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000 -1200 mg (Active Comparator): Sovaprevir 400 mg qd + ACH-3102 150 mg loading dose on Day 1, followed by 50 mg qd + RBV weight-based 1000-1200 mg qd for 12 weeks.
  Interventions: Drug: Sovaprevir; Drug: ACH-3102; Drug: Ribavirin
- Placebo (Placebo Comparator): Placebo for sovaprevir capsule qd + placebo for ACH-3102 150 mg loading dose on Day 1, followed by placebo for 50 mg qd + placebo for weight-based RBV qd for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sovaprevir — Nonstructural protein 3/4A protease inhibitor.
  Other Names: ACH-0141625
  Arms: Sovaprevir 200 milligrams (mg), ACH-3102 150/50 mg, RBV 1000-1200 mg; Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000 -1200 mg
Drug: ACH-3102 — Nonstructural protein 5A inhibitor.
  Arms: Sovaprevir 200 milligrams (mg), ACH-3102 150/50 mg, RBV 1000-1200 mg; Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000 -1200 mg
Drug: Ribavirin
  Arms: Sovaprevir 200 milligrams (mg), ACH-3102 150/50 mg, RBV 1000-1200 mg; Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000 -1200 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and efficacy of 12 weeks of treatment with sovaprevir, ACH-0143102, and ribavirin (RBV) in genotype-1 (GT-1), treatment-naive, hepatitis C virus (HCV) participants.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection.
* HCV GT-1.
* HCV ribonucleic acid > 10,000 international units/milliliter at screening.
* Female participants must be willing to use 2 effective methods of contraception, one of which must be a barrier method, during the dosing period and 6 months after the last dose of RBV. Females of childbearing potential must have a negative pregnancy test at screening and baseline.
* Male participants must be willing to use an effective barrier method of contraception throughout the dosing period and for 6 months.
* Signed and dated written informed consent form.
* Willing to participate in all study activities and all study requirements (including effective contraception) during the study period.
* Treatment-naïve participants were defined as those participants who have never received pegylated interferon, RBV, or a direct-acting anti-viral agent for the treatment of chronic HCV infection.
* A liver biopsy within the last 3 years without evidence of cirrhosis.

Exclusion Criteria:

* Body mass index > 36.0 kilograms/meter squared.
* Pregnant or nursing (lactating) female participants confirmed by a positive human chorionic gonadotropin laboratory test or contemplating pregnancy.
* Participation in any interventional clinical trial within 35 days prior to first study medication dose administration on Day 1.
* Known human immunodeficiency virus (HIV)-1 or HIV-2 infection/serology and/or positive hepatitis B surface antigen.
* Use of dietary supplements, grapefruit juice, herbal supplements, cytochrome P450 (CYP) 2C8 substrates, CYP3A4 inducers and inhibitors, P-glycoprotein inducers and substrates, organic-anion-transporting polypeptide inhibitors and substrates, and potent inducers of other CYP enzymes within 14 days prior to dosing through 7 days following completion of study medications.
* Clinically significant laboratory abnormality at screening (specified in protocol).
* Other forms of liver disease.
* History of severe or uncontrolled psychiatric disease.
* History of malignancy of any organ system, treated or untreated within the past 5 years.
* History of major organ transplantation.
* Use of bone marrow colony stimulating factor agents within 3 months prior to baseline.
* History of seizure disorder requiring ongoing medical therapy.
* History of known coagulopathy including hemophilia.
* History of hemoglobinopathy, including sickle cell anemia and thalassemia.
* History of immunologically mediated disease (specified in protocol).
* History of clinical evidence of significant chronic cardiac disease ( specified in protocol).
* Electrocardiogram with any clinically significant abnormality.
* Structural or functional cardiac abnormalities (specified in protocol).
* History of chronic obstructive pulmonary disease, emphysema, or other chronic lung disease.
* Participants currently abusing amphetamines, cocaine or opiates, or with ongoing alcohol abuse in the judgement of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 7 sites in the United States and 1 site in Canada between 07 May 2013 and 04 April 2014.
Pre-assignment Details: Participants were screened within 4 weeks (-28 to -1 days) before administration of the study drug. Participants who meet all eligibility criteria were instructed to arrive at the study center on baseline day.
Groups:
- Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg: Sovaprevir 200 milligrams (mg) once daily (qd) + ACH-3102 150 mg loading dose on Day 1, followed by 50 mg qd + ribavirin (RBV) weight-based 1000-1200mg qd for 12 weeks.
- Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg: Sovaprevir 400 mg qd + ACH-3102 150 mg loading dose on Day 1, followed by 50 mg qd + RBV weight-based 1000-1200 mg qd for 12 weeks.
Period: Overall Study
Arm/Group | Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Placebo
Started | 10 | 10 | 10
Completed | 8 | 10 | 10
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Non-compliance with Study Drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population for baseline characteristics was the safety population, defined as all randomized participants who received at least 1 dose of the study drug.
Groups:
- Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg: Sovaprevir 200 mg qd + ACH-3102 150 mg loading dose on Day 1, followed by 50 mg qd + RBV weight-based 1000-1200 mg qd for 12 weeks.
- Placebo: Placebo for sovaprevir capsule qd + placebo for ACH-3102 150 mg loading dose on Day 1 followed, by placebo for 50 mg qd + placebo for weight-based RBV qd for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 10 | 29
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (11.36) | 50.7 (8.51) | 53.8 (8.58) | 51.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 6 | 6 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 8 | 9 | 9 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 8 | 7 | 7 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kilograms] | 78.1 (15.02) | 81.5 (9.88) | 81.5 (11.9) | 80.2 (12.1)
Height [Mean (Standard Deviation); unit: Centimeters] | 170.1 (11.14) | 169.7 (9.76) | 175.6 (7.53) | 171.8 (9.66)

OUTCOME MEASURES:

1. Primary Outcome: Incidence Of Sustained Virologic Response 4 Weeks (SVR4) After The Completion Of Treatment
Description: Incidence of SVR4 after the completion of dosing, reported as hepatitis C virus (HCV) ribonucleic acid less than the lower limit of quantification, in participants who received active treatment (sovaprevir and ACH-0143102 in combination with RBV) as compared to those who received placebo.
Time Frame: Four weeks after the completion of treatment
Population: The analysis population for SVR4 was the full analysis (FA) set, defined as all randomized participants who received at least 1 dose of the study drug and had at least 1 baseline/post HCV RNA assessment. For this study, the FA set and the safety population were the same.
Measure: Number; unit: Percentage of participants with SVR4
Arm/Group | Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Percentage of participants with SVR4 | 50 | 70 | 0
Statistical Analysis 1: Comparison: Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg vs Placebo; Differences in proportions between Group 1 (sovaprevir 200 mg plus ACH-3102 150/50 mg plus RBV) and overall placebo (placebo from Group 1 and Group 2 combined) along with corresponding 95% confidence intervals for risk difference calculated using exact unconditional methods were obtained; Test type: Superiority or Other; Risk Difference (RD) = 50, 95% CI 2-sided [1.8 to 82.7]
Statistical Analysis 2: Comparison: Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg vs Placebo; Differences in proportions between Group 2 (sovaprevir 400 mg plus ACH-3102 150/50 mg plus RBV) and overall placebo (placebo from Group 1 and Group 2 combined) along with corresponding 95% confidence intervals for risk difference calculated using exact unconditional methods were obtained; Test type: Superiority or Other; Risk Difference (RD) = 70, 95% CI 2-sided [24.2 to 93.6]

2. Primary Outcome: Safety And Tolerability Of 12 Weeks Of Sovaprevir And ACH-3102 In Combination With RBV In GT-1 HCV Participants
Description: To determine the safety and tolerability of 12 weeks of sovaprevir/ACH-0143102/RBV treatment in participants with chronic genotype-1 (GT-1) HCV, the following criteria will be used: the number of participants with discontinuations due to adverse events (AEs), treatment-emergent Grade 3/Grade 4 (G3/G4) AEs, treatment-emergent G3/G4 laboratory abnormalities, and clinically significant electrocardiograms (ECGs).
Time Frame: 12 weeks
Population: The analysis population for safety and tolerability was the safety population, defined as all randomized participants who received at least 1 dose of study drug. For this study, the safety population and the FA set were the same.
Measure: Number; unit: participants
Groups:
- Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-2000 mg: Sovaprevir 400 mg qd + ACH-3102 150 mg loading dose on Day 1, followed by 50 mg qd + RBV weight-based 1000 -1200 mg qd for 12 weeks.
Arm/Group | Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-2000 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants
  Discontinuations due to AEs | 0 | 0 | 0
  Treatment Emergent G3/G4 AEs | 0 | 0 | 0
  Treatment Emergent G3/G4 Abnormalities | 3 | 2 | 0
  Clinically Significant ECGs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from enrollment into the study through end of treatment plus 24 weeks of follow-up.
Description: Treatment-emergent AEs were summarized.
Arm/Group | Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg (N=10) | Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg (N=10) | Placebo (N=10)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sovaprevir 200 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg (N=10) | Sovaprevir 400 mg, ACH-3102 150/50 mg, RBV 1000-1200 mg (N=10) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 4
Influenza like illness (General disorders) | 1 | 1 | 0
Irritability (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0/4 | 1/4 | 0/4
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/4 | 0/4 | 1/4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting/presenting a manuscript or materials relating to a Study to a publisher, reviewer, or outside person, the Institution shall provide to Sponsor a copy of all such manuscripts or materials, and Sponsor shall have thirty (30) days to review and comment. The Institution shall, upon Sponsor's request, further delay publication or presentation for a period of up to sixty (60) days to allow Sponsor to protect its interests in any Sponsor Inventions.